CLINICAL TRIAL: NCT03581383
Title: Implementation of Two Novel Interdisciplinary Care Models and the Impact on Hepatitis C Treatment Uptake, Completion, Sustained Virologic Response, and Retention in Care
Brief Title: Community Access, Retention in Care, and Engagement for Hepatitis C Treatment
Acronym: CARE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rosenau (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Jens Rosenau, Associate Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-0812-F2L
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Hep C; CARE-C; Kentucky
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: 3 Arms: Two intervention models plus a control group representing standard practice Arm 4: And intervention model to record patient experiences with telemedicine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Current Care Model (Control) (No Intervention): The Current Care Model will not have any intervention beyond the standard of care for Hepatitis C provided by an interdisciplinary team at the University of Kentucky.
- PREP-C Model (Experimental): The PREP-C care model will provide Hepatitis C care with the standard interdisciplinary team expanded by a social worker and a patient navigator team. The social worker/ patient navigator team will use the standardized Psychosocial Readiness Evaluation and Preparation for hepatitis C treatment (PREP-C) tool and will guide PREP-C related interventions to overcome barriers to HCV treatment uptake and completion.
  Interventions: Behavioral: PREP-C
- Modified ECHO Model (Experimental): The modified Extension for Community Healthcare Outcomes (ECHO) Model will provide patient care through collaboration of the expanded interdisciplinary team (including social worker patient navigator team) with community providers.
  Interventions: Behavioral: PREP-C; Behavioral: Modified ECHO
- Telemedicine Arm (Experimental): The telemedicine Model will track outcomes and record patient experiences with HCV management and treatment with telemedicine.
  Interventions: Behavioral: Patient Telemedicine Questionnaire

INTERVENTIONS:
Behavioral: PREP-C — The Psychosocial Readiness Evaluation and Preparation for Hepatitis C Treatment (PREP-C) is an interactive online tool that enables providers to provide a thorough assessment of a patient's psychosocial readiness to begin Hepatitis C treatment, and make a treatment plan to improve treatment readiness.
  Arms: Modified ECHO Model; PREP-C Model
Behavioral: Modified ECHO — The heart of the ECHO (Extension for Community Health Outcomes) model is its hub-and-spoke knowledge-sharing networks, led by expert teams who use multi-point videoconferencing to conduct virtual clinics with community providers. The key modification is one patient visit in the specialty center resulting in co-management of patients with data sharing.
  Arms: Modified ECHO Model
Behavioral: Patient Telemedicine Questionnaire — The patient questionnaire includes questions about patient experiences with telemedicine visits with providers
  Arms: Telemedicine Arm

SUMMARY:
The main goals of the CARE-C study are to demonstrate the effectiveness of HCV models of care in a rural state (A) to overcome barriers to HCV treatment uptake, (B) to increase retention in care, and (C) to broaden access to care. To achieve these goals the following two systems interventions will be separately implemented: (1) Implementation of the Psychosocial Readiness Evaluation and Preparation for hepatitis C treatment (PREP-C) and related standard of care best practice PREP-C related interventions facilitated by a social worker-patient navigator team, and (2) implementation of a modified ECHO model (with one patient visit at specialty center to include PREP-C and fibrosis assessment in contrast to standard ECHO model). To test the effectiveness of our two systems interventions 600 patients will be equally distributed into three study arms representing 3 care models: Arm 1: Current Care Model (management with current interdisciplinary team); Arm 2: PREP-C Model (management with expanded interdisciplinary team (social worker, patient navigator, PREP-C); and Arm 3: Modified ECHO Model (management with expanded team in collaboration with community providers). An additional Arm 4 was started January 2021 to follow subjects experience with HCV management and treatment via telemedicine.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) related complications (end-stage liver disease, liver cancer, and death) are increasing in the U.S., and extrapolated from U.S. data most of the estimated 49,200 patients with chronic hepatitis C in the state of Kentucky are untreated. In addition, the state of Kentucky is at the center of the rural opioid epidemic in the United States which has led to a dramatic increase in the transmission of hepatitis C virus (HCV) infection. HCV treatment uptake has been suboptimal in Kentucky despite the availability of highly effective, well-tolerated, timely limited treatment options due to multiple patient-, provider-, and system related barriers. Effective models of linkage to care, treatment, and retention in care are urgently needed to overcome the epidemiological challenges facing our rural state and put Kentucky on a path to planned elimination of HCV infection in the state. The demonstration of the effectiveness of new models of care in Kentucky which are appropriate to rural states will have great relevance and value to other states struggling with new HCV transmission and similar urgent need for effective models of linkage to care, treatment, and retention. Standardized care interventions expanding the reach of specialty providers (Project ECHO) and overcoming patient and provider related barriers to HCV treatment initiation (PREP-C assessment and interventions) have been evaluated, but the implementation of both models has been hampered by a lack of financial incentive, PREP-C has not been evaluated in rural populations, and the two models have never been used in conjunction.

The main goals of the study are to demonstrate the effectiveness of HCV models of care in a rural state (A) to overcome barriers to HCV treatment uptake, (B) to increase retention in care, and (C) to broaden access to care. To achieve these goals the following two systems interventions will be separately implemented: (1) Implementation of the Psychosocial Readiness Evaluation and Preparation for hepatitis C treatment (PREP-C) and related standard of care best practice PREP-C related interventions facilitated by a social worker-patient navigator team, and (2) implementation of a modified ECHO model (with one patient visit at specialty center to include PREP-C and fibrosis assessment in contrast to standard ECHO model). To test the effectiveness of our two systems interventions up to 1000 participants will be distributed into four study arms representing 4 care models: Arm 1, Current Care Model (management with current interdisciplinary team);arm 2, PREP-C Model (management with expanded interdisciplinary team (social worker, patient navigator, PREP-C); arm 3, Modified ECHO Model (management with expanded team in collaboration with community providers); and Arm 4, current Telemedicine care model (management with current interdisciplinary team).

The specific aims are:

Aim 1: To compare HCV treatment uptake within 12 months after the first clinic visit (time of enrollment) in all Arms 1, 2, and 3. It is hypothesized that (A) treatment uptake will be higher in Arms 2 (PREP-C model) and 3 (modified ECHO model) as compared to Arm 1 (current care model) as a result of overcoming patient level treatment barriers (such as ongoing substance use, psychiatric instability, non-compliance, loss to follow up) facilitated by implementation of the PREP-C assessment, PREP-C related interventions, and assistance of the social worker-patient navigator team, and (B) treatment uptake in Arm 3 will be non-inferior to Arm 2.

Aim 2: To compare HCV treatment outcomes (treatment completion and sustained virologic response, SVR12) in all arms 1, 2, and 3. It is hypothesized that treatment completion and SVR12 in arms 2 and 3 will be noninferior to arm 1 due PREP-C enhancement, even though expected additional patients who start treatment in Arms 2 and 3 are expected to have less favorable treatment readiness scores prior to PREP-C interventions due to higher rates of treatment uptake as hypothesized in Aim 1.

Aim 3: To compare retention in care in all 3 arms for patients who do not start treatment (within 12 months after initial appointment). It is hypothesized that retention in care will be higher in arms 2 and 3 due to implementation of PREP-C assessment and interventions, and the support through the patient navigator.

Aim 4: To record the treatment uptake and analyze patient experiences with telemedicine appointments in Arm 4, the telemedicine arm.

ELIGIBILITY:
Inclusion Criteria:

* First office visit for hepatitis C management
* Referred either (a) to the Hepatology Outpatient Clinic at the University of Kentucky in Lexington, Kentucky or (b) to a local community provider who can provide comprehensive care for HCV including HCV treatment in collaboration with the University of Kentucky as a spoke of the ECHO program
* Age 18 years and older

Exclusion Criteria:

* Life expectancy less than one year
* Less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
HCV treatment initiation | 12 months
  The overall number of patients who have started HCV treatment by month12 after the first clinic visit will be divided by the number of patients enrolled and presented as a percentage of participants per group.
HCV treatment completion | 12 months
  The number of patients who have completed HCV treatment will be divided by the number of patients who have started treatment and presented as a percentage of participants per group.
Sustained Virologic Response (SVR) | 12 weeks from treatment completion
  The number of patients who achieve sustained virologic response (negative HCV RNA 12 weeks after completion of HCV treatment) will be divided by the number of patients who have started treatment and presented as a percentage of participants per group.

SECONDARY OUTCOMES:
Missed clinic visits | 18 months
  The total number of missed clinic visits will be counted for each group. Data will be presented as the number of missed visits divided by the number of total visits scheduled and presented as a percentage of total clinic appointments.
Clinic visit consistency | 18 months
  This outcome will measure the number of participants attending clinical visits with less than six month intervals between visits. Data will be presented as the number of participants maintaining an appointment interval less than six months divided by the total number of participants.
Gaps in clinical care | 18 months
  The average time between clinical appointments will be calculated between groups. Data will be presented as the mean amount of time +/- SEM.
Appointment adherence | 18 months
  This outcome will measure the number of clinical appointments the participant attended compared to the number of appointments they were scheduled to attend. Data presented as the ratio of attended/scheduled appointments
Visit frequency within a twelve month period | 18 months
  This outcome will track the number of participants attending two or more clinical appointments in a 12 month period with at least 3 months between visits. Data will be presented as the ratio of participants in each group attending multiple visits compared to the total number of participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rosenau, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No